CLINICAL TRIAL: NCT00039845
Title: fMRI Languages Studies In Young Children
Brief Title: MRI Language Studies in Young Children
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020223; 02-N-0223
Record Dates: First submitted 2002-06-12; First posted 2002-06-13 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-04-20

CONDITIONS: Healthy
Keywords: Brain; Imaging; Pediatrics; Mapping; Development; fMRI; Children; Language; Healthy Volunteer; HV; Normal Control
MeSH Terms: conditions — Language

SUMMARY:
This study will use magnetic resonance imaging (MRI) to investigate language function in children-that is, how language skills such as naming objects, understanding spoken language and reading are organized in the brain. The study focuses on children between 4 and 7 years old. Children 8 to 12 years old and adults will be studied before the younger children to test study paradigms appropriate for pre-literate children. The results of this study will help evaluate the usefulness of MRI in identifying language function and location and may improve the treatment of children with seizures.

Right-handed, native English-speaking adults and children between 4 and 12 years of age may be eligible for this study. Candidates will be screened with a routine neurological examination. Children will also undergo neuropsychological testing (standard tests of language, memory, perception and attention) either at the screening visit or at a later time. Parents will fill out a form to identify children with attention deficit and hyperactivity disorders. These children will be excluded form the study.

All participants will undergo MRI scanning of the brain while performing a task designed to test a language skill, such as identifying a picture or listening to or reading a word. The MRI detects changes in blood properties in the areas of the brain that perform each task. Before the MRI, children will be rehearsed for the tests and will have a session in the scanner to know what to expect and feel more at ease during the actual test. The time in the MRI machine is usually between 15 and 20 minutes, but will be no more than 40 minutes for children 8 to 12 years old, and not more than 20 minutes for younger children. Children may be requested to have up to five MRI sessions to test different brain functions or confirm findings.

...

DETAILED DESCRIPTION:
This protocol aims to develop paradigms to identify the neural networks that underlie language processing in pre/early literate children. These studies are designed to test the hypothesis that language networks are strongly lateralized and regionally specific in children younger than eight. The study extends our investigations of paradigm development and language network organization in adults and older children (8-12) to the 4-7 year age group. Word reading, object naming, and auditory comprehension paradigms will be adapted for children 4-7 years old. Paradigm stimuli will be devised from pilot data obtained under protocol 01-N-181. Paradigms will be piloted in adults and older children (8-12 years) before young child studies (4-7 years) and will employ the 1.5 and 3T scanners. Paradigms will be designed to overcome limitations in previous studies: monitoring performance in the scanner, using 3T and event related designs to improve signal to noise and allow data analysis in relation to task item response, and improve motion correction, using language neutral control conditions, and using paradigms appropriate for pre-literate children. Data will be analyzed on an individual basis with AFNI and group analysis with SPM 99 using random effect analysis to identify brain regions associated with task performance. These paradigms will be used as language probes for other protocols designed to study the effect of acute and chronic disease states (e.g. stroke and epilepsy) on the plasticity of neuronal organization in language networks. In order to compare two non-invasive language mapping modes, we will perform magnetoencephalography with auditory category and description decision tasks.

ELIGIBILITY:
* INCLUSION CRITERIA:

Right handed (Edinburgh Handedness Inventory).

Native English speaker.

Adults and older children (8-12 years) will be recruited to pilot paradigms. Younger children, aged 4-7 years, are the principal subject of the study.

EXCLUSION CRITERIA:

Medical contraindications to MRI procedures (e.g. pacemakers, cochlear devices, surgical clips, etc).

Technical contraindications to MRI procedures (e.g. no braces (distort image data)).

History of neurologic or psychiatric disease or a learning or attentional disorder.

School performance one year below grade level.

CNS active medications.

Pregnancy.

Claustrophobia.

Inability to comply with the protocol.

Volunteers will also be asked if they have a history of dry or irritated eyes and informed this may increase the risk of eye irritation and discomfort in the 3T scanner.

Ages: 4 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 180
Dates: Start 2002-06-07; Study Completion 2009-04-20

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Barnes PD. Imaging of the central nervous system in pediatrics and adolescence. Pediatr Clin North Am. 1992 Aug;39(4):743-76. doi: 10.1016/s0031-3955(16)38374-2. PMID 1635805
- [Background] Benson RR, FitzGerald DB, LeSueur LL, Kennedy DN, Kwong KK, Buchbinder BR, Davis TL, Weisskoff RM, Talavage TM, Logan WJ, Cosgrove GR, Belliveau JW, Rosen BR. Language dominance determined by whole brain functional MRI in patients with brain lesions. Neurology. 1999 Mar 10;52(4):798-809. doi: 10.1212/wnl.52.4.798. PMID 10078731
- [Background] Binder JR, Rao SM, Hammeke TA, Frost JA, Bandettini PA, Jesmanowicz A, Hyde JS. Lateralized human brain language systems demonstrated by task subtraction functional magnetic resonance imaging. Arch Neurol. 1995 Jun;52(6):593-601. doi: 10.1001/archneur.1995.00540300067015. PMID 7763208